CLINICAL TRIAL: NCT03682055
Title: Phase 1/2a Open Label, Multicenter Clinical Trial of a Novel Small Molecule EBNA1 Inhibitor, VK 2019, in Patients With Epstein Barr Virus Positive Nasopharyngeal Cancer, With Pharmacokinetic and Pharmacodynamic Correlative Studies
Brief Title: Phase 1/2a Study of VK-2019 in Patients With Epstein-Barr Virus (EBV)-Positive Nasopharyngeal Carcinoma (NPC)
Status: Terminated | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: Lack of efficacy
Sponsor: Cullinan Therapeutics Inc. (Industry)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: VK-2019-001
Record Dates: First submitted 2018-09-20; First posted 2018-09-24 (Actual); Results first posted 2023-08-15 (Actual); Last update posted 2023-08-15 (Actual); Status verified 2023-07

CONDITIONS: Nasopharyngeal Carcinoma; Nasopharyngeal Cancer
Keywords: Epstein-Barr Virus; Nasopharyngeal Carcinoma; NPC; EBV; EBNA1 inhibitor; VK-2019; Nasopharynx cancer; Nasopharynx carcinoma
MeSH Terms: conditions — Nasopharyngeal Carcinoma; Nasopharyngeal Neoplasms; Epstein-Barr Virus Infections

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- Phase 1 Dose Escalation (Accelerated Titration) (Experimental): VK-2019 QD in Accelerated Titration dose escalation cohorts enrolling EBV+ NPC
  Interventions: Drug: VK-2019
- Phase 1 Dose Escalation (Rolling Six) (Experimental): VK-2019 QD in Rolling Six dose escalation cohorts enrolling EBV+ NPC.
  Interventions: Drug: VK-2019
- Phase 1 Dose Expansion(s) (Experimental): VK-2019 QD in expansion cohorts that may be opened at doses that meet pre-specified criteria for clinical and/or biological activity.
  Interventions: Drug: VK-2019
- Phase 2a Dose Expansion(s) (Experimental): VK-2019 QD in expansion cohorts that may be opened at doses that meet pre-specified efficacy criteria in Phase 1 Dose Escalation cohorts.
  Interventions: Drug: VK-2019

INTERVENTIONS:
Drug: VK-2019 — EBNA1 inhibitor

SUMMARY:
VK-2019-001 is a 1/2a trial of the oral EBNA-1 targeting agent VK-2019 in patients with EBV-positive recurrent or metastatic NPC to determine the Maximum Tolerated Dose (MTD) and Recommended Phase 2 Dose (RP2D), as well as to evaluate the PK profile of VK-2019.

DETAILED DESCRIPTION:
This is a Phase 1/2a, open-label, multicenter, first-in-human trial to evaluate the safety and tolerability, PK, PD, and preliminary efficacy of VK-2019 in patients with EBV-positive NPC.

This trial is divided into three parts: Phase 1 Dose Escalation, Phase 1 Dose Expansion, and Phase 2s Dose Expansion.

The objectives of the dose escalation part are to determine the safety, tolerability, MTD, recommended Phase 2 dose (RP2D), and to evaluate the anti-tumor activity of orally administered VK-2019 monotherapy. Additional objectives are to determine the pharmacokinetic (PK) profile of VK-2019.

VK-2019 will be dosed once daily (QD).

ELIGIBILITY:
Inclusion Criteria:

1. Informed consent obtained prior to any protocol mandated assessment.
2. Age ≥ 18.
3. Either loco regionally recurrent or metastatic EBV positive nasopharyngeal carcinoma not amenable to curative treatment. EBV positivity is defined as high EBV viral load in plasma (> 4000 genomes per µg plasma DNA) and/or biopsy tissue positive for EBV.
4. Prior palliative radiation must have been completed at least 2 weeks prior to study Cycle 1 Day 0.
5. Prior anti cancer systemic treatment must have been completed greater than 4 weeks prior to study Cycle 1 Day 0.
6. Toxicities related to prior anti-cancer therapy must have returned to Grade 1 or less. Peripheral neuropathy must be Grade 2 or less. Chronic but stable toxicities Grade > 1 (e.g., dysphasia, G tube dependence, etc.) may be allowed after agreement between the Investigator and Sponsor.
7. For the dose expansion phase only: Patients must have RECIST v1.1 measurable disease, defined as at least one lesion that can be accurately measured in at least one dimension (longest diameter to be recorded for non nodal lesions and short axis for nodal lesions) as ≥ 10 mM with spiral CT scan, MRI, or calipers by clinical exam.
8. ECOG performance status score of ≤ 2 at study entry.
9. Absolute neutrophil count > 1500/µL (stable off any growth factor within 1 week of study drug administration).
10. Hemoglobin > 9g/dL (transfusion to achieve this level is permitted).
11. Platelet count > 75 x 103/ µL (transfusion to achieve this level is NOT permitted).
12. Serum aspartate transaminase (AST) and serum alanine transaminase (ALT) ≤ 2.5 x upper limit of normal (ULN).
13. Total serum bilirubin ≤ 1.5 x ULN.
14. Serum creatinine ≤ 1.5 x ULN or creatinine clearance ≥ 50 mL/min as calculated per Cockcroft Gault equation.
15. Urinary protein < 2+ by dipstick. If dipstick ≥ 2+, then a 24 hour urine collection can be done and the patient may enter only if urinary protein is < 1 g/24 hour.
16. Sexually active patients must agree to utilize birth control method during the study and for 18 weeks after the study is concluded, using effective birth control methods as defined in https://www.cdc.gov/reproductivehealth/unintendedpregnancy/pdf/contraceptive_methods_508.pdf.
17. Willingness and ability to comply with the study scheduled visits, treatment plans, laboratory tests and other procedures.

Exclusion Criteria:

1. Severe or active symptomatic cardiopulmonary diseases (unstable angina and/or congestive heart failure or peripheral vascular disease within the last 12 months; chronic obstructive pulmonary disease exacerbation other respiratory illness requiring hospitalization) or clinically significant psychiatric disorders; patients with effectively treated conditions (eg, stenting for CAD) are eligible.
2. Metastatic disease with active central nervous system (CNS) involvement, defined as parenchymal brain involvement. Patients with cranial nerve or base of skull involvement without the above are eligible; Patients with CNS metastases stable 1 month following focal treatment with radiation are eligible.
3. Concurrent treatment with systemic cancer directed therapy including complementary, alternative, herbal or nutritional supplement based treatments whose purpose is for anti cancer effect.
4. Positive for human immunodeficiency virus (HIV) are not excluded from this study, but HIV positive patients must have:

   * A stable regimen of highly active anti retroviral therapy (HAART)
   * No requirement for concurrent antibiotics or antifungal agents for the prevention of opportunistic infections
   * A CD4 count above 250 cells/mcL and an undetectable HIV viral load on standard PCR based test
5. Serious uncontrolled medical disorder or active infection which would, in the opinion of the Investigator, impair the ability of the subject to receive protocol therapy or whose control may be jeopardized by the complications of this therapy.
6. Currently taking drugs that inhibit or induce OATP1B1 or OATP1B3 within 5 half lives of that agent. Examples are included in Appendix 2.
7. Have received a prior organ allograft or allogeneic bone marrow transplant.
8. Current non prescription drug or alcohol dependence.
9. For all female patients, pregnancy or breastfeeding.
10. All female patients with reproductive potential must have a negative pregnancy test (serum or urine) prior to enrollment.
11. Other severe acute or chronic medical or psychiatric condition or laboratory abnormality that may increase the risk associated with study participation or study drug administration, or may interfere with the interpretation of study results, or in the judgment of the investigator would make the patient inappropriate for entry into the study.
12. Corrected QT by Fridericia's formula (QTcF) of > 470 ms.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 14 (Actual)
Dates: Start 2019-04-04 (Actual); Primary Completion 2020-06-23 (Actual); Study Completion 2020-08-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: A. Dimitrios Colevas, MD, Study Chair — Stanford Cancer Institute
Locations (6):
- United States (2):
  - Stanford University, School of Medicine, Stanford Cancer Institute, Stanford, California
  - The University of Texas - MD Anderson Cancer Center, Houston, Texas
- Sun Yat Sen University Cancer Center, Guangzhou, Guangdong, China
- Institut Gustave Roussy, Villejuif, France
- Hong Kong University - Queen Mary Hospital, Hong Kong, Hong Kong
- National Cancer Centre Singapore, Singapore, Singapore

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Young LS. Epstein-Barr virus at 50-future perspectives. Chin J Cancer. 2014 Nov;33(11):527-8. doi: 10.5732/cjc.014.10208. PMID 25367333
- [Background] Young LS, Dawson CW. Epstein-Barr virus and nasopharyngeal carcinoma. Chin J Cancer. 2014 Dec;33(12):581-90. doi: 10.5732/cjc.014.10197. Epub 2014 Nov 21. PMID 25418193
- [Background] Tsao SW, Tsang CM, Lo KW. Epstein-Barr virus infection and nasopharyngeal carcinoma. Philos Trans R Soc Lond B Biol Sci. 2017 Oct 19;372(1732):20160270. doi: 10.1098/rstb.2016.0270. PMID 28893937

RESULTS

PARTICIPANT FLOW:
Groups:
- Cohort 1 (Phase 1 Accelerated Titration): 60 mg QD
- Cohort 2 (Phase 1 Accelerated Titration): 120 mg QD
- Cohort 3 (Phase 1 Accelerated Titration): 230 mg QD
- Cohort 4 (Phase 1 Accelerated Titration): 460 mg QD
- Cohort 5 (Phase 1 Accelerated Titration): 920 mg QD
- Cohort 6 (Phase 1 Rolling 6): 1800 mg QD
Period: Overall Study
Arm/Group | Cohort 1 (Phase 1 Accelerated Titration) | Cohort 2 (Phase 1 Accelerated Titration) | Cohort 3 (Phase 1 Accelerated Titration) | Cohort 4 (Phase 1 Accelerated Titration) | Cohort 5 (Phase 1 Accelerated Titration) | Cohort 6 (Phase 1 Rolling 6)
Started | 1 | 2 | 1 | 2 | 1 | 7
Completed | 0 | 0 | 0 | 0 | 0 | 0
Not Completed | 1 | 2 | 1 | 2 | 1 | 7
Not completed — Lack of Efficacy | 1 | 2 | 1 | 2 | 1 | 3
Not completed — Withdrawal by Subject | 0 | 0 | 0 | 0 | 0 | 1
Not completed — Termination of Study by Sponsor | 0 | 0 | 0 | 0 | 0 | 3

BASELINE CHARACTERISTICS:
Groups:
- Cohort 6 (Phase 1 Accelerated Titration): 1800 mg QD
- Total: Total of all reporting groups
Arm/Group | Cohort 1 (Phase 1 Accelerated Titration) | Cohort 2 (Phase 1 Accelerated Titration) | Cohort 3 (Phase 1 Accelerated Titration) | Cohort 4 (Phase 1 Accelerated Titration) | Cohort 5 (Phase 1 Accelerated Titration) | Cohort 6 (Phase 1 Accelerated Titration) | Total
Number analyzed (Participants) | 1 | 2 | 1 | 2 | 1 | 7 | 14
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Between 18 and 65 years | 1 | 1 | 1 | 1 | 1 | 7 | 12
  >=65 years | 0 | 1 | 0 | 1 | 0 | 0 | 2
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1 | 1 | 0 | 0 | 0 | 1 | 3
  Male | 0 | 1 | 1 | 2 | 1 | 6 | 11
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Asian | 1 | 2 | 1 | 1 | 1 | 3 | 9
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Black or African American | 0 | 0 | 0 | 0 | 0 | 0 | 0
  White | 0 | 0 | 0 | 1 | 0 | 0 | 1
  More than one race | 0 | 0 | 0 | 0 | 0 | 1 | 1
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 3 | 3
Region of Enrollment [Number; unit: participants]
  Hong Kong | 0 | 0 | 0 | 0 | 1 | 2 | 3
  United States | 1 | 2 | 1 | 2 | 0 | 2 | 8
  France | 0 | 0 | 0 | 0 | 0 | 3 | 3

OUTCOME MEASURES:

1. Primary Outcome: All Cohorts: The Frequency, Severity, and Duration of AEs and DLTs, AEs Leading to Discontinuation, and AEs Leading to Death.
Time Frame: 24 months
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort 1 (Phase 1 Accelerated Titration) | Cohort 2 (Phase 1 Accelerated Titration) | Cohort 3 (Phase 1 Accelerated Titration) | Cohort 4 (Phase 1 Accelerated Titration) | Cohort 5 (Phase 1 Accelerated Titration) | Cohort 6 (Phase 1 Rolling 6)
Number analyzed (Participants) | 1 | 2 | 1 | 2 | 1 | 7
Participants
  Experienced a DLT | 0 | 0 | 0 | 0 | 0 | 0
  Experienced a treatment related AE leading to discontinuation | 0 | 0 | 0 | 0 | 0 | 0
  Experienced a treatment-related AE leading to death | 0 | 0 | 0 | 0 | 0 | 0
  Experienced an AE | 1 | 2 | 1 | 2 | 1 | 7

2. Secondary Outcome: Phase 1 Dose Escalation and Dose Expansion Cohorts: ORR
Time Frame: 24 months
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort 1 (Phase 1 Accelerated Titration) | Cohort 2 (Phase 1 Accelerated Titration) | Cohort 3 (Phase 1 Accelerated Titration) | Cohort 4 (Phase 1 Accelerated Titration) | Cohort 5 (Phase 1 Accelerated Titration) | Cohort 6 (Phase 1 Rolling 6)
Number analyzed (Participants) | 1 | 1 | 1 | 2 | 1 | 3
Participants
  Stable Disease | 1 | 0 | 0 | 0 | 1 | 1
  Progressive Disease | 0 | 0 | 1 | 2 | 0 | 2
  Partial Response | 0 | 0 | 0 | 0 | 0 | 0
  Complete Response | 0 | 0 | 0 | 0 | 0 | 0
  Missing / Not Evaluable | 0 | 1 | 0 | 0 | 0 | 0

ADVERSE EVENTS:
Time Frame: 1 year, 8 months
Arm/Group | Cohort 1 (Phase 1 Accelerated Titration) | Cohort 2 (Phase 1 Accelerated Titration) | Cohort 3 (Phase 1 Accelerated Titration) | Cohort 4 (Phase 1 Accelerated Titration) | Cohort 5 (Phase 1 Accelerated Titration) | Cohort 6 (Phase 1 Rolling 6)
All-Cause Mortality (participants affected / at risk) | 0/1 | 1/2 | 0/1 | 0/2 | 0/1 | 0/7
Serious Adverse Events (participants affected / at risk) | 0/1 | 2/2 | 0/1 | 0/2 | 1/1 | 3/7
Other Adverse Events (participants affected / at risk) | 1/1 | 2/2 | 1/1 | 2/2 | 1/1 | 7/7
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Cohort 1 (Phase 1 Accelerated Titration) (N=1) | Cohort 2 (Phase 1 Accelerated Titration) (N=2) | Cohort 3 (Phase 1 Accelerated Titration) (N=1) | Cohort 4 (Phase 1 Accelerated Titration) (N=2) | Cohort 5 (Phase 1 Accelerated Titration) (N=1) | Cohort 6 (Phase 1 Rolling 6) (N=7)
Malignant neoplasm progression (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Tumour Pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Pleural Effusion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Tracheal Stenosis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Urinary Tract Infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Gastrostomy tube site complication (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Cohort 1 (Phase 1 Accelerated Titration) (N=1) | Cohort 2 (Phase 1 Accelerated Titration) (N=2) | Cohort 3 (Phase 1 Accelerated Titration) (N=1) | Cohort 4 (Phase 1 Accelerated Titration) (N=2) | Cohort 5 (Phase 1 Accelerated Titration) (N=1) | Cohort 6 (Phase 1 Rolling 6) (N=7)
Not Reported (Social circumstances) | 1 (1) | 2 (2) | 1 (1) | 2 (2) | 1 (1) | 7 (7) — Since no clinical and PD activity could be demonstrated, the sponsor decided to prematurely end the study and listings of AEs by subject were not generated.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2019-10-15): https://cdn.clinicaltrials.gov/large-docs/55/NCT03682055/Prot_000.pdf
  • Statistical Analysis Plan (2020-11-12): https://cdn.clinicaltrials.gov/large-docs/55/NCT03682055/SAP_001.pdf